CLINICAL TRIAL: NCT01288378
Title: Empirical Versus Pre-emptive (Diagnostic-driven) Antifungal Therapy of Patients Treated for Haematological Malignancies or Receiving an Allogeneic Stem Cell Transplant. A Therapeutic Open Label Phase III Strategy Study of the EORTC Infectious Diseases and Leukemia Groups
Brief Title: Empirical Versus Preemptive Antifungal Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EORTC-65091-06093; 2010-020814-27 (EudraCT Number); MK-0991-070 (Other: Merck (MSD))
Record Dates: First submitted 2011-02-01; First posted 2011-02-02 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Fungal Infection; Leukemia; Myelodysplastic Syndromes
Keywords: fungal infection; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; recurrent adult acute myeloid leukemia; untreated adult acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with del(5q); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); secondary acute myeloid leukemia
MeSH Terms: conditions — Mycoses; Leukemia; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Congenital Abnormalities | interventions — Caspofungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Empirical (Active Comparator): Empirical approach (fever driven) for starting antifungal therapy
  Interventions: Drug: caspofungin acetate
- Pre-emptive (Experimental): Pre-emptive approach (diagnostic driven) for starting antifungal therapy
  Interventions: Drug: caspofungin acetate

INTERVENTIONS:
Drug: caspofungin acetate — intravenous route, at a 70 mg loading dose on day 1 of antifungal therapy, followed by 50 mg once a day thereafter.

SUMMARY:
RATIONALE: Caspofungin acetate may be effective in treating fungal infections in patients with acute myeloid leukemia or myelodysplastic syndrome who are receiving treatment for their cancer. It is not yet known whether caspofungin acetate is more effective when treatment starts after development of a fever or after the infection is shown in laboratory test, chest x-ray, or CT scan.

PURPOSE: This randomized phase III trial is studying the best time to start caspofungin acetate therapy in treating patients with acute myeloid leukemia or myelodysplastic syndrome that is newly diagnosed or in first relapse.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare empirical approach (i.e., fever driven) versus preemptive approach (i.e., diagnostic driven), for starting antifungal therapy with caspofungin acetate, in patients with acute myeloid leukemia or myelodysplastic syndrome who are starting chemotherapy (for attaining remission induction) or myeloablation (to prepare for an allogeneic hematopoietic stem cell transplantation) for newly diagnosed disease or disease in first relapse.

Secondary

* To evaluate clinical validity and utility of a standardized Aspergillus PCR assay.
* To evaluate clinical validity and utility of beta-D-glucan.
* To determine the occurrence of single nucleotide polymorphisms (SNPs) and the predictive value of SNPs for identifying patients at higher risk of developing invasive fungal infection.

OUTLINE: This is a multicenter study. Patients are stratified according to institution, prior allogeneic stem cell transplantation (yes vs no), and type of air flow (laminar air flow vs high-efficiency particulate air). Patients are randomized to 1 of 2 treatment arms.

* Arm A (Empirical approach): Patients start caspofungin acetate treatment when one of the following criteria are met:

  * Presence of unexplained persistent fever refractory to 4 full days of broad-spectrum antibacterial therapy with any of the following regimens either alone or in combination with an aminoglycoside or a glycopeptide:

    * Ceftazidime
    * Cefepime
    * Piperacillin/tazobactam
    * Imipenem-cilastatin
    * Meropenem
  * New fever occurring > 2 days after resolution of a first fever while continuing broad-spectrum antibacterial therapy as defined above for which no obvious cause has been documented and fungal infection cannot be excluded Patients receive caspofungin acetate IV once daily. Treatment continues until neutrophil recovers.
* Arm B (Preemptive approach): Patients start caspofungin acetate treatment when at least one of the following criteria* are met:

  * Single plasma or serum galactomannan ELISA with index > 0.5
  * New pulmonary infiltrate on chest x-ray and IFD cannot be readily excluded
  * New dense well-circumscribed lesions with or without a halo sign, on a CT scan, consistent with IFD
  * Aspergillus sp. recovered by culture from sputum Patients receive caspofungin acetate IV once daily. Treatment continues until neutrophil recovers.

NOTE: *These criteria are not sufficient to warrant preemptive caspofungin acetate therapy: skin lesions evocative of IFD, sinusitis or orbititis, hepatosplenic abscesses (hypodensities on CT scan), or unexplained persistent fever for more than 7 days or recurrent fever whatever its duration.

All patients undergo blood sample collection periodically for the detection of galactomannan and beta-D-glucan and for the detection of single nucleotide polymorphisms. Some patients undergo blood sample collection for the detection of Aspergillus via PCR. An economic evaluation is performed for cost-effectiveness analysis.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS)

  * Newly diagnosed disease or disease in first relapse after hematological remission lasting for a minimum of 6 months AND meets one of the following criteria:

    * Starting remission-induction chemotherapy within 3 days prior to study randomization
    * Starting myeloablative conditioning regimen to prepare for a first allogeneic hematopoietic stem cell transplantation within 3 days prior to study randomization
* Planning a hospital admission for the duration of the neutropenic phase (ANC < 0.5 x 10^9 /L)
* Planning to receive oral or intravenous fluconazole for Candida prophylaxis at a dose of 400 mg/day

  * Fluconazole is discontinued during caspofungin acetate administration
* No previous or current history of proven or probable invasive fungal disease (IFD)

PATIENT CHARACTERISTICS:

* See Disease Characteristics
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients muse use effective contraception during and for at least 3 months after completion of study therapy
* No current clinical diagnosis of pneumonia
* No serious, uncontrolled, concomitant disease or comorbidity that, in the opinion of the investigator, may compromise adherence to the study protocol
* No history of allergy or any adverse reaction to echinocandin drugs (i.e., caspofungin acetate, micafungin, or anidulafungin)
* No hypersensitivity to caspofungin active substance or to any of the excipients
* No inadequately treated infection
* No documented HIV infection
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* No history of liver cirrhosis or severe hepatic insufficiency (i.e., Child Pugh Class C, D, or E)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent participation on another clinical trial using an investigational drug for infectious diseases
* No other concurrent systemic antifungal therapy (oral or intravenous)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Actual)
Dates: Start 2012-03; Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Overall survival at 42 days after randomization | 6 weeks after randomization

SECONDARY OUTCOMES:
Overall survival at 84 days after randomization | 12 weeks after randomization
Development of proven or probable invasive fungal disease (IFD) during the 42 and 84 days following randomization | during 84 days after randomization
Proper management according to allocated treatment arm (i.e., appropriate administration of caspofungin acetate in compliance to protocol, and compliance to the treatment strategy) during the 42 and 84 days after randomization | during 84 days after randomization
Survival-free of fungal infection during the 42 and 84 days following randomization | during 84 days after randomization
Safety (adverse event [AE] and serious adverse event [SAE]) as assessed by CTCAE criteria v4.0 | during 84 days after randomization
Number of days under caspofungin treatment or under another antifungal treatment administered after caspofungin (evaluation will be done at day 42 and day 84 after randomization) | at day 42 and day 84 after randomization
Costs related to the strategy for initiating and monitoring antifungal treatment during the 42 and 84 days following randomization | during 84 days after randomization

CONTACTS AND LOCATIONS:
Locations (16):
- Belgium (5):
  - A.Z. St. Jan, Bruges
  - Cliniques Universitaires Saint-Luc, Brussels
  - Hôpitaux Universitaires Bordet-Erasme - Institut Jules Bordet, Brussels
  - U.Z. Gasthuisberg, Leuven
  - C.H.U. Sart-Tilman, Liège
- Masaryk University, Brno, Czechia
- France (6):
  - CHU de Caen - Hopital Cote de Nacre, Caen
  - C.H.U. Henri Mondor AP-HP, Créteil
  - CHRU de Lille - Hopital Hurie, Lille
  - CHU de Limoges - Hopital Dupuytren, Limoges
  - Hopital Universitaire Hautepierre, Strasbourg
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Universitaetsklinikum Wuerzburg - Medizinische Klinik und Poliklinik II, Würzburg
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands
- National Cancer Institute, Bratislava, Slovakia

REFERENCES:
- [Derived] Maertens J, Lodewyck T, Donnelly JP, Chantepie S, Robin C, Blijlevens N, Turlure P, Selleslag D, Baron F, Aoun M, Heinz WJ, Bertz H, Racil Z, Vandercam B, Drgona L, Coiteux V, Llorente CC, Schaefer-Prokop C, Paesmans M, Ameye L, Meert L, Cheung KJ, Hepler DA, Loeffler J, Barnes R, Marchetti O, Verweij P, Lamoth F, Bochud PY, Schwarzinger M, Cordonnier C; Infectious Diseases Group and the Acute Leukemia Group of the European Organization for Research and Treatment of Cancer. Empiric vs Preemptive Antifungal Strategy in High-Risk Neutropenic Patients on Fluconazole Prophylaxis: A Randomized Trial of the European Organization for Research and Treatment of Cancer. Clin Infect Dis. 2023 Feb 18;76(4):674-682. doi: 10.1093/cid/ciac623. PMID 35906831